CLINICAL TRIAL: NCT06720025
Title: A Phase 3 Study to Compare the Efficacy and Safety of SAL-0951 With Recombinant Human Erythropoietin Injection in Anemic Patients With Chronic Kidney Disease Receiving Maintenance Hemodialysis <Switch / Maintenance Study>
Brief Title: Study of SAL-0951 Compared to Recombinant Human Erythropoietin in Anemic Patients Receiving Maintenance Hemodialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Salubris Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAL0951A302
Record Dates: First submitted 2024-12-02; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Anemia
Keywords: Anemia; Renal Insufficiency; Chronic Dialyses; Renal Dialyses; Renal Hemodialysis; Hematinic; Hematopoietic Agents; Erythropoiesis Stimulating Agents; Enarodustat; rHuEPO
MeSH Terms: conditions — Anemia; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAL-0951 tablets (Experimental): initial phase：4mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: SAL-0951 tablets
- rHuEPO injection (Active Comparator): Initial based on the original rHuEPO dose adjust the dose based on hemoglobin concentration level every 4 weeks
  Interventions: Drug: rHuEPO injection

INTERVENTIONS:
Drug: SAL-0951 tablets — initial phase：4mg QD subsequent phase：1mg～8mg QD，adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: SAL-0951 group
  Arms: SAL-0951 tablets
Drug: rHuEPO injection — Initial based on the original rHuEPO dose adjust the dose based on hemoglobin concentration level every 4 weeks
  Other Names: rHuEPO group
  Arms: rHuEPO injection

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of SAL-0951 in Chinese patients undergoing maintenance hemodialysis with chronic kidney disease and anemia，who are receiving stable treatment with erythropoietic stimulants (ESAs).

DETAILED DESCRIPTION:
A randomized, open-label, rHuEPO positive-controlled, parallel-design multicenter clinical trial is used to evaluate the efficacy and safety of SAL-0951 in maintenance hemodialysis patients with anemia in CKD who were stable on ESAs. It is planned to enroll 100 subjects and eligible subjects screened are assigned 1:1 to the test arm and the control arm for a 24-week treatment to verify that the efficacy of SAL-0951 in the treatment of renal anemia in hemodialysis patients is non-inferior to that of rHuEPO and to verify the long-term safety of investigational drug in the treatment of renal anemia by comparing the difference in mean Hb levels between the two arms at weeks 20, 22, and 24 after treatment.

The study is mainly divided into four stages: screening period (2 weeks before administration), initial treatment period (4 weeks), maintenance treatment period (20 weeks), and safe follow-up period (2 weeks), requiring a total of 12 visits. This study included the 24th week visit as the end of treatment visit (EOT) and the 26th week as the end of study visit (EOS). Subjects who withdrew early are required to complete the research procedure for week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Patients receiving hemodialysis (including hemodiafiltration) consistently three times a week for at least 12 weeks before Scr Visit 1.Dialysis is performed through autologous arteriovenous fistula or graft fistula (artificial blood vessel) or permanent tunnel catheter (central venous catheter with cuff).
2. Patients with TSAT*1 >20% or ferritin >75 μg/L at Scr Visit 1

   *1: If serum iron values are invalid values, TSAT values shall also be handled as invalid values and re-test will be performed (For patients with ferritin >75 μg/L, there is no need for re-test).
3. Patients who have continued to receive the treatment with the same ESAs (rHuEPO or DA) for at least 4 weeks before Scr Visit 1
4. Patients receiving ESAs for at least 2 weeks before Scr Visit 1 satisfying a) and c), or b) and c) below

   1. Patients receiving rHuEPO once to three times weekly, and at a total weekly dose of ≥750 IU and ≤9,000 IU
   2. Patients receiving DA once weekly, and at a dose of 10 µg, 20 μg or 30 μg
   3. Patients receiving ESAs at a constant total weekly dose for 2 weeks before Scr Visit 1
5. Patients who have received the same ESAs as received in most recent week before Scr Visit 1 during the period between Scr Visit 1 and the day before Week 0 at the same total dose and dosing frequency a week*1

   *1: If ESAs is administered once weekly on the third dialysis day (Friday, if dialysis is performed, for instance, on Monday, Wednesday, and Friday), ESAs administration on the third dialysis day immediately before Week 0 will not be performed.
6. Patients with pre-dialysis Hb levels measured after the maximum interdialytic interval at Scr Visit 1 and Scr Visit 2 (1 week after the start of observation) of ≥95 g/L and <120 g/L and a difference (in absolute value) between Scr Visit 1 and Scr Visit 2 of ≤10 g/L
7. Weight 45 to 100 kg

Exclusion Criteria:

1. Patients with poorly controlled hypertension (e.g., systolic blood pressure ≥180 mmHg and diastolic blood pressure ≥110 mmHg at Scr Visit 1 and Scr Visit 2)
2. Patients with severe hepatobiliary disease (e.g., AST or ALT >2.5x upper limit of normal value at Scr Visit 1, hepatic cirrhosis, total bilirubin 1.5x upper limit of normal value at Scr Visit 1
3. Patients with congestive heart failure (NYHA Class III or IV) or unstable angina
4. Patients who have developed myocardial infarction, cerebral infarction (excluding asymptomatic cerebral infarction), or venous thromboembolism (pulmonary embolism or deep vein thrombosis or dialysis vascular pathway thrombosis or occlusion) during the period between 24 weeks before Scr Visit 1 and the registration to the treatment period
5. Patients who will undergo an ophthalmological procedure (photocoagulation therapy or vitreous surgery) for the treatment of diabetic retinopathy, diabetic macular edema, or age- related macular degeneration during the period between Scr Visit 1 and the end of the study
6. Patients who have undergone erythrocyte transfusion during the period between 12 weeks before Scr Visit 1 and the registration to the treatment period (according to clinical treatment indications, transfusions of blood products that do not contain red blood cells may be excluded, such as plasma, albumin, etc.)
7. Patients who have received protein anabolic hormones, testosterone enanthate, or mepitiostane during the period between 12 weeks before Scr Visit 1 and the registration to the treatment period
8. Patients with severe hyperparathyroidism (e.g., intact-PTH ≥500 pg/mL at Scr Visit 1)
9. Patients with severe infections (such as active pulmonary tuberculosis, fungal infections, etc.), systemic hematological diseases (such as myelodysplastic syndrome, aplastic anemia, abnormal hemoglobin disease, etc.) or hemolytic anemia, or patients with anemia caused by bleeding disorders (such as gastrointestinal bleeding, etc.)
10. Except for glomerulonephritis, anemia patients suspected to be caused by non infectious chronic inflammatory diseases such as systemic lupus erythematosus, rheumatoid arthritis, celiac disease, etc.
11. Patients with malignancy (including hematological malignancy), except for tumors determined to be cured or in remission for 5 years, skin basal cell or squamous cell carcinoma that has undergone radical resection, or in situ carcinoma of any part
12. Patients with a history of severe drug allergies, such as anaphylactic shock or allergies to rHuEPO or other HIF-PHI
13. Patients with current or previous history of drug dependence or alcohol dependence within the past 2 years
14. Patients who have received another investigational product (or study drug), have received treatment with an investigational device (or study device), or have participated in clinical research involving intervention (medical action beyond the scope of ordinary medical practice intended for research purposes) and received treatment during the period between 12 weeks before Scr Visit 1 and the registration to the treatment period
15. Patients who have previously participated in a clinical study of SAL-0951 and received the investigational product (active drug)
16. Patients who are pregnant, lactating, or may be pregnant (the possibility of pregnancy cannot be ruled out by the PI or the SI based on the results of pregnancy test at Scr Visit 1
17. Female patients of childbearing potential who have not agreed to use appropriate contraception methods from the time of signing of informed consent to the end of the study, or male patients who have not agreed to use appropriate contraception methods*1 from the start of study treatment to the end of the study

    *1 appropriate contraception methods Effective contraceptive methods include transdermal patches, oral medication, implantable or injectable contraceptives, abstinence or birth control surgery
18. Diagnosed as polycystic kidney disease
19. Positive for any of the following: human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), or anti hepatitis C virus antibodies (anti HCV Ab), or confirmed syphilis requiring treatment
20. Received treatment with SAL-0951 or other HIF-PH inhibitors within the first 8 weeks of randomization
21. Any other medical condition that, in the opinion of the investigator, could pose a safety risk to the subject in this study, could confound efficacy or safety assessment, or could interfere with the subject's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Difference in mean hemoglobin (Hb) level between arms during the evaluation period after treatment (non-inferiority margin: -10 g/L) | weeks 20, 22, and 24
  Hb levels during the evaluation period after treatment are defined as the mean value of Hb levels at weeks 20, 22, and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Ph.D, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No